CLINICAL TRIAL: NCT06045845
Title: The Effects of Beetroot Supplementation and Habitual Dietary Nitrate Intake on Exercise Performance in Collegiate Female Rowing Athletes
Brief Title: Effects of Beet Juice and Diet in Female Rowers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Jessica Provost, Principal Investigator, Doctoral Candidate, Graduate Teaching Assistant, University of Kansas Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: STUDY00150492
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Dietary Habits; Nitrates; Exercise
Keywords: dietary nitrate; beetroot juice; sex differences; exercise; performance; muscle
MeSH Terms: conditions — Feeding Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Beet Juice First (Experimental): First Test: Beet Juice / Second Test: Placebo
  Interventions: Dietary Supplement: Beet Juice; Dietary Supplement: Placebo
- Placebo Beet Juice First (Experimental): First Test: Placebo / Second Test: Beet Juice
  Interventions: Dietary Supplement: Beet Juice; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beet Juice — 70 milliliter (70mL) standard Beet Juice (Beet It Sport Shot) consumed 2.5 hours before exercise test
Dietary Supplement: Placebo — 70mL placebo Beet Juice (Beet It Sport Shot with nitrate removed) consumed 2.5 hours before exercise test

SUMMARY:
The purpose of this study is to determine the effects of nitrate-rich beetroot juice supplementation on exercise performance in female rowers when accounting for habitual vegetable nitrate consumption.

DETAILED DESCRIPTION:
The objective is to use a stratified block randomization, double-blind crossover trial to test rowing ergometer exercise performance after drinking a beetroot juice supplement and compare it to the same test after consuming a placebo (a nitrate-free version of the beetroot juice supplement) in a convenience sample of athletes from a single Division 1-A collegiate women's rowing team.

Before testing, the participants' habitual vegetable nitrate consumption will be assessed from their report of foods consumed in the past 24 hours. Estimates of dietary nitrate intake will be calculated from the quantity of vegetables consumed and used to determine whether dietary nitrate intake influences the efficacy of the beetroot juice supplement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Athletes currently on the university's rowing team

Exclusion Criteria:

* Injuries or medical conditions that prevent participation in their team's rowing training program
* Diagnosis of stage 2 iron deficiency
* Unable to consume beet juice for any reason

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Rowing Test Time | Recorded immediately upon completion of each of the 4 500-meter intervals during rowing time trial tests on day 7 and day 14.
  Time (seconds) to complete 500-meter rowing time trial tests.
Rowing Test Perceived Exertion | Recorded immediately upon completion of each of the 4 500-meter intervals during rowing time trial tests on day 7 and day 14.
  Rating of perceived exertion reported by participant during rowing time trial tests. The Borg Scale is used, in which participants choose a number between 6 ("Rest") and 20 ("Maximal Effort") to indicate their perceived exertion at the completion of each 500-meter segment.
Rowing Test Peak Heart Rate | Recorded during each of the 4 500-meter intervals during rowing time trial tests on day 7 and day 14.
  Maximum heart rate (beats per minute) during 500-meter rowing time trial tests. The Maximum is the single highest heart rate recorded during that 500-meter interval.
Rowing Test Average Heart Rate | Recorded during each of the 4 500-meter intervals during rowing time trial tests on day 7 and day 14.
  Mean heart rate (beets per minute) during 500-meter rowing time trial tests.
Rowing Test Peak Power Output | Recorded during each of the 4 500-meter intervals during rowing time trial tests on day 7 and day 14.
  Maximum power (watts) during 500-meter rowing time trial tests
Rowing Test Average Power Output | Recorded during each of the 4 500-meter intervals during rowing time trial tests on day 7 and day 14.
  Mean power (watts) during 500-meter rowing time trial tests
Dietary Nitrate Habitual Consumption Amount | Collected after each rowing time trial test for the preceding 24-hour period (day 6 and day 13). Means determined in post-testing analysis.
  Mean vegetable nitrate consumption (mg/day) from two different self-administered 24-hour dietary recalls (ASA24).
Dietary Nitrate Habitual Consumption Category | Collected after each rowing time trial test for the preceding 24-hour period (day 6 and day 13). Median and categories determined in post-testing analysis.
  Categorization of Dietary Nitrate Habitual Consumption Amount. The median of all participants' Amounts will be determined to categorize each participant as "high" (above median) or "low (below median).

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A Provost, MS, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Rowing Boathouse, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Upon completion of the testing protocol, all data analysis will be conducted using only using the de-identified participant identification numbers. There is no plan to share individual participant data with other researchers.